CLINICAL TRIAL: NCT04365972
Title: Attention Bias Modification for Reducing Health Anxiety During the Coronavirus Pandemic: An Open Pilot Trial
Brief Title: Attention Bias Modification for Reducing Health Anxiety During the Coronavirus Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Prof. Yair Bar-Haim, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAU-COVID-19
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-delivered attention bias modification (ABM) (Experimental): A home-delivered ABM comprised of 5 sessions using a variant of the dot-probe task in which the target probe always replaces neutral rather than threat (health-related) stimuli to induce diversion of attention away from threat.
  Interventions: Behavioral: Attention Bias Modification (ABM)

INTERVENTIONS:
Behavioral: Attention Bias Modification (ABM) — A home-delivered version of ABM will be administered in this open trial. ABM will be comprised of 5 sessions with a variation of the dot-probe task in which the target probe always replaces the neutral stimuli to induce diversion of attention away from threat. This condition was found effective in reducing anxiety symptoms.

SUMMARY:
The outbreak of the 2019 Coronavirus (COVID-19) pandemic is a major stressor leading to increased levels of anxiety, and specifically, an excessive fear of being infected and affected by the disease among major parts of the population. At the same time, the access to mental health services is limited due to the lockdown policy applied in many countries worldwide, warranting the development of home-delivered interventions aimed at reducing stress and anxiety symptoms. Attention Bias modification (ABM) has been found to be an efficacious computerized intervention to reduce anxiety symptoms. In this open pilot trial, participants reporting on elevated levels of health anxiety concerning the COVID-19 epidemic will receive one session of ABM over 5 consecutive days (5 sessions total). Symptoms of health anxiety, state anxiety, generalized anxiety, and depression will be measured at baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more symptoms (out of 7) reported in the COVID-19 anxiety inventory with a score of 4 or 5.
* Fluent Hebrew
* Having a PC computer at home with internet access

Exclusion Criteria:

* A diagnosis of dyslexia or other reading disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the total score of a novel COVID-19 anxiety inventory | up to 2 days pre-treatment and 1-2 days post-treatment
  The COVID-19 anxiety inventory is a self-report questionnaire screening for concerns and fears regarding COVID-19 contagion. The Inventory consists of 6 items. Scores can range from 6 to 30, with higher scores denoting higher symptom severity.

SECONDARY OUTCOMES:
Change from baseline of the total score of the Health Anxiety Inventory | up to 2 days pre-treatment and 1-2 days post-treatment
  The Health Anxiety Inventory (HAI) is a validated self-report measure assessing health anxiety. Total score can range from 0 to 42, with higher scores denoting higher symptom severity
Change from baseline of the total score of the State Anxiety Inventory | up to 2 days pre-treatment and 1-2 days post-treatment
  The State Anxiety Inventory is a validated self-report measure for state anxiety. Total score can range from 20 to 80, with higher scores denoting higher levels of state anxiety.
Change from Baseline of the total score of the PHQ-9 | up to 2 days pre-treatment and 1-2 days post-treatment
  The PHQ-9 is a 9-item self-report scale for depression symptoms. Scores can range from 0 to 27, with higher scores reflecting more symptoms of depression.
Change from Baseline of the total score of the GAD-7 | up to 2 days pre-treatment and 1-2 days post-treatment
  The GAD-7 is a 7-item self-report scale for generalized anxiety symptoms. Scores can range from 0 to 21, with higher scores reflecting more symptoms of generalized anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No